CLINICAL TRIAL: NCT00835211
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of TEVA and Aventis Pharmaceuticals (DDAVP®) 0.2 mg Desmopressin Acetate Tablets in Healthy Adult Subjects Following a 0.8 mg Dose Under Fasting Conditions
Brief Title: Desmopressin Acetate 0.2 mg Tablets, Fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA04887
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Desmopressin Acetate 0.2 mg Tablets
- 2 (Active Comparator)
  Interventions: Drug: DDAVP® 0.2 mg Tablets

INTERVENTIONS:
Drug: Desmopressin Acetate 0.2 mg Tablets — 4 x 0.2 mg, single-dose fasting
  Arms: 1
Drug: DDAVP® 0.2 mg Tablets — 4 x 0.2 mg, single-dose fasting
  Arms: 2

SUMMARY:
The objective of this study was to compare the single-dose relative bioavailability of TEVA and Aventis Pharmaceuticals (DDAVP®) 0.2 mg desmopressin acetate tablets following a 0.8 mg dose under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult non-smoker (for at least 3 months) or light smoking (less than 10 cigarettes per day for at least 3 months) male or female subjects, 18-55 years of age;
* Weighing at least 60 kg for males and 52 kg for females;
* Subjects who had a body mass index (BMI) less than 30;
* Medically healthy subjects with clinically normal laboratory profiles and ECGs;

Females of childbearing potential should have either been sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or have been using one of the following acceptable birth control methods:

* surgically sterile (tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum. Proof was required for the hysterectomy and oophorectomy;
* IUD in place for at least 3 months;
* barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the first dose and throughout the study;
* surgical sterilization of the partner (vasectomy for 6 months minimum);
* hormonal contraceptives for at least 3 months prior to the first dose of the study.

Other birth control methods were deemed acceptable. Postmenopausal women with amenorrhea for at least 2 years were eligible.

* Voluntarily consent to participate in the study.

Exclusion Criteria:

* Female subjects who were pregnant or lactating.
* Subjects who had been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.
* Any clinically significant illness within 4 weeks prior to dosing.
* Subjects with any medical condition requiring regular treatment with prescription drugs.
* The use of any pharmacological agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to the first dose.
* Subjects who, through completion of the study, would have donated in excess of: 500 mL of blood and/or plasma in 14 days; 1500 mL of blood and/or plasma in 180 days; 2500 mL of blood and/or plasma in 1 year.
* Subjects who had donated plasma within 30 days prior to the first dose.
* Subjects who ahd participated in another clinical trial within 30 days prior to the first dose.
* Subjects who did not tolerate venipuncture.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.

In addition, the history or presence of:

* hypersensitivity or idiosyncratic reaction to desmopressin or any other synthetic anti-diuretic hormones;
* type IIB von Willebrand's disease;
* personal or family bleeding disorder;
* alcoholism or drug abuse within the past year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2003-07; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, M.D., Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Sercives, Saint-Laurent, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Desmopressin Acetate: Desmopressin Acetate 4 x 0.2 mg Tablet (test) dosed in first period followed by DDAVP® 4 x 0.2 mg Tablet (reference) dosed in second period
- DDAVP®: DDAVP® 4 x 0.2 mg Tablet (reference) dosed in first period followed by Desmopressin Acetate 4 x 0.2 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Desmopressin Acetate | DDAVP®
Started | 24 | 24
Completed | 24 | 23
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout: 7 Days
Arm/Group | Desmopressin Acetate | DDAVP®
Started | 24 | 23
Completed | 21 | 22
Not Completed | 3 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Desmopressin Acetate | DDAVP®
Started | 21 | 22
Completed | 21 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desmopressin Acetate | DDAVP® | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 12 | 18 | 30
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 22 | 20 | 42
  Hispanic | 2 | 2 | 4
  Black | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 12 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Desmopressin Acetate: Desmopressin Acetate 4 x 0.2 mg Tablet (test) dosed in either period
- DDAVP®: DDAVP® 4 x 0.2 mg Tablet (reference) dosed in either period
Arm/Group | Desmopressin Acetate | DDAVP®
Number analyzed (Participants) | 43 | 43
pg/mL | 78.102 (52.5437) | 82.888 (64.2238)
Statistical Analysis 1: Comparison: Desmopressin Acetate vs DDAVP®; Test type: Non-Inferiority or Equivalence — Analyses of Variance (ANOVA) were performed on the log-transformed AUC0-t, AUCinf and Cmax. These analyses were performed using the SAS® procedure; Test/Ref Ratio of LS Means x 100 = 97.5, 90% CI [87.8 to 108.3] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUCinf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUCinf
Time Frame: Blood samples collected over 12 hour period
Population: AUC0-inf could not be estimated for one subject in the reference arm.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Desmopressin Acetate | DDAVP®
Number analyzed (Participants) | 43 | 42
pg*h/mL | 266.62 (169.435) | 286.34 (199.268)
Statistical Analysis 1: Comparison: Desmopressin Acetate vs DDAVP®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 95.6, 90% CI [86.9 to 105.2] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 12 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Desmopressin Acetate | DDAVP®
Number analyzed (Participants) | 43 | 43
pg*h/mL | 252.85 (162.914) | 268.02 (188.907)
Statistical Analysis 1: Comparison: Desmopressin Acetate vs DDAVP®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 96.5, 90% CI [87.7 to 106.1] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.